CLINICAL TRIAL: NCT07216768
Title: ADAPT: Approach to Dance for Autism
Acronym: ADAPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Ballet Academy East (Unknown)
Responsible Party: Principal Investigator, Alexander Kolevzon, Director of Child and Adolescent Psychiatry for the Mount Sinai Health System; Clinical Director of the Seaver Autism Center, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY-25-00779
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Ballet; Recreational dance; Autism Spectrum Disorder; motor coordination; social skills
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

STUDY DESIGN:
Intervention Model Description: Participants will participate in 12 weeks of recreational ballet classes following the established Ballet For All Kids curriculum. Participants will have weekly 45 minute classes with videos covering moves taught in class that are to be watched 3x/week. In class, participation and balance scales will be used to evaluate motor function. Parents or guardians will complete questionnaires at baseline, 6 weeks, and completion of the program. This study is a waitlist control model, where one group will complete surveys in the fall while not receiving the intervention, and again in the Spring while taking the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 - Classes in fall (Experimental): Participants randomly assigned to cohort 1 will begin classes in fall 2025. Parents/guardians will complete surveys just one time over the 12 week intervention
  Interventions: Behavioral: Ballet Class
- Cohort 2 - Classes in spring (Experimental): This cohort is a waitlist control. Parents/guardians will complete all surveys during the fall while their children do not receive the intervention. They will then receive the intervention in the spring and surveys will be completed again.
  Interventions: Behavioral: Ballet Class

INTERVENTIONS:
Behavioral: Ballet Class — Participants will attend weekly ballet classes following either Level 1 or Level 2 Ballet For All Kids (BFAK) curriculum.

SUMMARY:
It is well documented that motor impairments are associated with a diagnosis of autism spectrum disorder (ASD). Yet, appropriate therapies are scarce. Dance has been shown to not only promote fine and gross motor skills, but also psychological well-being, cognition, and social participation in neurotypical dancers. Little research has been conducted to gauge if these benefits translate to those with ASD. Ballet for all Kids (BFAK) is a recreational dance program that has been teaching ballet to children with ASD for over a decade, but has yet to be empirically studied. This study expands on the goals of former STUDY 24-00144, Approach to Dance for Autism (ADAPT), NCT06424366, to elucidate the impact of participation in a recreational dance program on children with ASD.

DETAILED DESCRIPTION:
The researchers aim to expand upon the pilot randomized trial (STUDY-24-00144) using BFAK's curriculum and structure to elucidate the impact of a recreational ballet program on the motor function and psychological, social, and behavioral skills of children with ASD. For the primary objective, the researchers hypothesize that after 12 weeks of participation in BFAK, children with ASD will improve their motor function. For the secondary objectives, the researchers hypothesize that after 12 weeks of participation in BFAK, children with ASD will improve their behavior and mood. This is a single site, randomized trial with 32 individuals diagnosed with ASD.

Participants will be placed in either Level 1 or Level 2 based on prior experience with BFAK. Participants returning from our pilot study will be placed into Level 2 at the discretion of the program coordinators, and all newly recruited participants will be placed in Level 1. BFAK ballet classes will begin in September and run for 45 minutes once a week for the intervention group. The waitlist control group will begin classes in January for 45 minutes once a week, ending in March 2026.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years age
* understand English or Spanish
* Autism Spectrum Disorder diagnosis
* not currently taking ballet class

Exclusion Criteria:

- none

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-05-03 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
Change in Developmental Coordination Disorder Questionnaire (DCDQ) | baseline, week 6,and week 12
  The change in scores on the DCDQ at baseline and weeks 6 and 12 of the BFAK program.
  The DCDQ is a 15 item questionnaire designed to screen for coordination challenges in children from 5 to 15 years old and has long been used in children with ASD. It comprises 3 subscales: (1) Control during movement (scale 9-45), (2) Fine Motor/Handwriting (scale 11-55), and (3) General Coordination (scale 10-50).
  Scores are calculated by weighting the domains as follows: (Control during movement/30) + (Fine Motor/Handwriting/20) + (General Coordination/25) = TOTAL, reported as a range from 15-75. Higher scores indicate better coordination.
  For Children Ages 5 years 0 months to 7 years 11 months: 5-46 indication of DCD or suspect DCD; 47-75 probably not DCD
  For Children Ages 8 yrs 0 mos to 9 yrs 11 mos: 15-55 indication of DCD or suspect DCD; 56-75 probably not DCD
  For Children Ages 10 yrs 0 mos to 15 yrs: 15-57 indication of DCD or suspect DCD; 58-75 probably not DCD
Change in Pediatric Balance Scale | baseline and week 12
  The difference in participants' scores on the Pediatric Balance scale at baseline and week 12.
  The Pediatric Balance Scale is a 14-item questionnaire that prompts children to complete certain movements such as standing unsupported, turning 360 degrees, and retrieving an object from the floor. Completion of movements are scored on a scale from 0 to 4. Full scale is scored 0-56, with higher scores corresponding to more advanced motor skills.
Change in Movement Assessment Battery for Children. | baseline and weeks12
  The difference in participants' scores on the Movement Assessment Battery for Children (MABC) at baseline and week 12.
  The MABC is a standardized tool used to identify and describe motor impairments in children. It assesses fine and gross motor skills across everyday movement domains, and is commonly used for diagnosing Developmental Coordination Disorder (DCD) and related difficulties. The MABC is divided into three domains: (1) Manual Dexterity (0-15), (2) Aiming & Catching (0-10), (3) Balance (0-15).
  Full scale is scored from 0-40 as a sum of the three domains. A higher total score indicates greater motor difficulty/impairment. Lower scores indicate better motor competence.

SECONDARY OUTCOMES:
Aberrant Behavior Checklist (ABC) | baseline, week 6, week 12
  The difference in participants' scores on self-reports of the Aberrant Behavior Checklist (ABC) at baseline, week and completion of the BFAK program.
  The ABC is a 58-item scale designed to assess the impact of treatment on various presentations and behaviors of developmental disorders and has been widely used in children with ASD. The ABC is divided into five main subscales: Irritability/Agitation/Crying (0-45), Lethargy/Social Withdrawal (0-48), Stereotypic Behavior (0-21), Hyperactivity/Noncompliance (0-48), and Inappropriate Speech (0-12). Total score ranges from 0 to 174. Higher scores indicate more severe problems.
Swanson, Nolan and Pelham (SNAP-IV) | baseline, week 6, week 12
  The difference in SNAP-IV scores on self-reports at baseline and week 6, completion.
  The SNAP-IV is a DSM-based symptom rating scale commonly used to assess ADHD symptoms (Inattention; Hyperactivity/Impulsivity) with an optional Oppositional Defiant Disorder (ODD) domain. Total score ranges from 0 to 78 on the 26-item version (higher scores indicate greater symptom severity). The SNAP-IV is divided into three subscales: Inattention (0-27), Hyperactivity/Impulsivity (0-27), and Oppositional Defiant (0-24). If using only the 18 ADHD items, the ADHD Total ranges from 0 to 54. Higher scores indicate more severe problems.
Number of classes attended | baseline, week 6, week 12
  The difference in active participation across attended classes as measured by in-house designed rubrics completed by volunteers at each class.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Adler, BSc, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan or need for this data to be shared at this time. However we are collecting parent/guardian consent for future use of de-identified data.